CLINICAL TRIAL: NCT03440983
Title: OSS-IRM: Optimization of MRI Sequences in Healthy Volunteers
Acronym: OSS-IRM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2011-A01531-40
Record Dates: First submitted 2013-04-08; First posted 2018-02-22 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-02

CONDITIONS: Healthy
Keywords: optimize the imaging protocols; validate technical parameters in healthy volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MRI data acquiring in healthy volunteers (Experimental): MRI data acquiring in healthy volonteers
  Interventions: Device: MRI data acquiring in healthy volunteers

INTERVENTIONS:
Device: MRI data acquiring in healthy volunteers — The quality of the images, cartographies or spectres will be compared to standard acquisitions. This evaluation will be based on qualitative visual criteria assessed by expert radiologists or on quantitative criteria assessed by data processing tools

SUMMARY:
Using MRI, many technical parameters can be changed to optimize the diagnostic quality of the examination. The study is interventionnal because healthy volunteers are not supposed to have an MRI exam.

The primary objective of this study is to optimize the imaging protocols and to validate the choice of the technical parameters in healthy volunteers.

The quality of the images, cartographies or spectres will be compared to standard acquisitions. This evaluation will be based on qualitative visual criteria assessed by expert radiologists or on quantitative criteria assessed by data processing tools.

DETAILED DESCRIPTION:
Using MRI, many technical parameters (sequence, parameters in the sequence, reconstruction method, etc.) can be changed to optimize the diagnostic quality of the examination.

The primary objective of this study is to optimize the imaging protocols and to validate the choice of the technical parameters in healthy volunteers.

The quality of the images, cartographies or spectres will be compared to standard acquisitions. This evaluation will be based on qualitative visual criteria assessed by expert radiologists or on quantitative criteria assessed by data processing tools.

Prospective, single-center, observational MRI study A screening visit is planned to check the inclusion/non inclusion criteria followed by an imaging visit during which the MRI examination will be performed.

Theses 2 visits are scheduled at the subject's convenience. The number of participations to the study is limited to 5 per year per subject.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject,
* Aged 18 or above

Exclusion Criteria:

* Patient with any surgical clip, external clips, or any other ferromagnetic device, that is contraindicated for use in MRI
* Claustrophobic patient
* Pregnancy
* Breastfeeding
* Patients subject to major legal protection (safeguarding justice, guardianship, trusteeship), persons deprived of liberty
* No healthcare insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2013-04; Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
MRI data acquisition : quality of the images, cartographies or spectres | 0.5 day
  The quality of the images, cartographies or spectres will be compared to standard acquisitions. This evaluation will be based on qualitative visual criteria assessed by expert radiologists or on quantitative criteria assessed by data processing tools

CONTACTS AND LOCATIONS:
Locations (1):
- Radiology Department CHU de Rennes, Rennes, France